CLINICAL TRIAL: NCT04420806
Title: Effects of Three Months of COVID-19 Lockdown Induced Deconditioning After 13 Months of High Intensity Exercise Training in Early Postmenopausal Women
Brief Title: Effects of COVID-19 Lockdown in Exercising Early Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ER_ACTLIFE_FU
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Exercise; Detraining; Muscle Weakness; Muscle Atrophy
MeSH Terms: conditions — Motor Activity; Muscle Weakness; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: One exercise versus one control group
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are unaware of participants group status and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIT-exercise (Active Comparator): 13 months of high intensity endurance and resistance exercise - 3 months of exercise break
  Interventions: Other: HIT-exercise
- control (Sham Comparator): no exercise intervention that affect the present study outcomes
  Interventions: Other: Sham intervention

INTERVENTIONS:
Other: HIT-exercise — 13 months of high intensity endurance and resistance exercise, 3x 45 min/week - 3 months of COVID-19 induced exercise break
  Arms: HIT-exercise
Other: Sham intervention — Types of exercise (flexibility, relaxation) that did not affect the present outcomes
  Arms: control

SUMMARY:
While "conditioning" by exercise training has been widely evaluated, the available literature on "passive deconditioning" (i.e. forced deconditioning) is predominately limited to studies with or with almost complete mechanical and/or metabolic immobilization/sedation of the respective functional system (e.g. paralysis, bedriddenness). Vice versa, the effects of moderately long interruptions of dedicated types of exercise while maintaining everyday activity are rarely addressed. However, this topic is of high relevance, e.g. considering that breaks of health-related exercise programs due to increased family/occupational stress, vacation or temporary orthopedic limitation are rather frequent in everyday life. In the present project we aimed to determine the effects of 3 months of physical deconditioning due to COVID-19 induced lockdown after 13 month of high intensity endurance and resistance exercise in early postmenopausal women on parameters related to health and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* (early)postmenopausal women, ( normal menopause, 1-5 years post)
* Osteopenia and osteoporosis (Bone Mineral Density <-1.0 SD T-Score)

Exclusion Criteria:

* BMD <-4.0 SD T-Score
* Prevalent clinical, low-trauma fractures
* Diseases and drugs with relevant effects on bone and muscle metabolism (e.g. glucocorticoids >7.5 mg/d or bisphosphonate therapy); individual case assessment
* Diseases and drugs with relevant effects on cardiometabolic risk factors (e.g. severe hypertension with corresponding medical therapy); individual case assessment
* Severe cardiovascular events (e.g. stroke, coronary infarction) in the past.
* Other conditions, diseases that exclude exercise training or testing

Ages: 48 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — early postmenopausal status
Enrollment: 21 (Actual)
Dates: Start 2020-03-14 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Body composition | From intervention end to 3 months FU
  Body composition as determined by Dual-Energy x-Ray Absorptiometry

SECONDARY OUTCOMES:
Hip-/Leg extension strength | From intervention end to 3 months FU
  Hip-/Leg extension strength as determined by an isokinetic leg press
Metabolic Syndrome | From intervention end to 3 months FU
  cardio-metabolic risk factors summarized in the Metabolic Syndrome Z-Score according to the definition of the International Diabetes Federation
Bone Mineral Density (BMD) | From intervention end to 3 months FU
  BMD at the lumbar spine and total hip as determined by Dual Energy x-Ray Absorptiometry
Menopausal symptoms | From intervention end to 3 months FU
  Menopausal symptoms as determined by the "Menopausal Rating Scale" (MRS) with a scale from 0 (no complaints) to 4 (very serious complaints).
Back and joint pain | From intervention end to 3 months FU
  Back and joint pain as determined by a standardized pain questionnaire with a scale from 0 (never) to 7 (permanent) for pain frequency or 0 (no pain) to 7 (extremely) for pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hettchen, MSc, Principal Investigator — Institute of Medical Physics, Friedrich-Alexander University Erlangen-Nürnberg
Locations (1):
- Institute of Medical Physics, Friedrich-Alexanden University Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kemmler W, Hettchen M, Kohl M, Murphy M, Bragonzoni L, Julin M, Risto T, von Stengel S. Detraining Effects on Musculoskeletal Parameters in Early Postmenopausal Osteopenic Women: 3-Month Follow-Up of the Randomized Controlled ACTLIFE Study. Calcif Tissue Int. 2021 Jul;109(1):1-11. doi: 10.1007/s00223-021-00829-0. Epub 2021 Mar 12. PMID 33712920